CLINICAL TRIAL: NCT03484078
Title: Effect of Vibration on Muscle Properties, Physical Activity and Balance in Children with Cerebral Palsy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Collaborators: Emory University (Other)
Responsible Party: Principal Investigator, Christopher Modlesky, Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STUDY00004873
Record Dates: First submitted 2018-03-13; First posted 2018-03-30 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy, Spastic
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: Children with CP will be randomly assigned to a vibration or a placebo group.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Vibration Platform (Experimental): The vibration group will stand on a platform that emits a mild vibration 10 minutes per day for 6 months. There will also be a 6 month no-treatment period.
  Interventions: Device: Vibration Platform
- Placebo Platform (Placebo Comparator): The placebo group will stand on a placebo platform 10 minutes per day for 6 months. There will also be a 6 month no-treatment period.
  Interventions: Device: Placebo Platform

INTERVENTIONS:
Device: Vibration Platform — The vibration platform will emit a mild vibration when the participant stands on it 10 minutes per day for 6 months.
  Arms: Vibration Platform
Device: Placebo Platform — The placebo platform will not vibrate when the participant stands on it 10 minutes per day for 6 months.
  Arms: Placebo Platform

SUMMARY:
The aim of the 6-month randomized controlled trial, with 6-month no treatment follow-up, is to examine the effects of low-magnitude vibration on muscle, physical activity, and balance in children with spastic cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a movement disorder that affects over 800,000 people in the U.S. Due to the limited mobility associated with the disorder, individuals with CP have an increased risk of chronic diseases, such as cardiovascular disease, diabetes mellitus and osteoporosis, compared to the general population. Therefore, identifying treatment strategies is of utmost importance. The aim of this study is to examine the acute and chronic effects of low-magnitude vibration on muscle, physical activity, and balance in children with CP. Fat concentration and muscle will be assessed using imaging techniques. Physical activity will be assessed using activity monitors. Balance will be assessed using clinical and biomechanical tests. Children with CP will be tested at five time points: baseline, 1 and 6 months after standing on a vibration platform daily 10 minutes per day, 1 and 6 months post treatment (7 months and 12 months from baseline, respectively). The findings from the proposed study will help us determine if vibration shows promise as a treatment for the impaired mobility, lower physical activity and higher risk of chronic disease in individuals with CP.

ELIGIBILITY:
Inclusion Criteria:

* Spastic cerebral palsy
* Independent ambulator without an assistive device (Gross Motor Function Classification System level I or II)

Exclusion Criteria:

* Prior fractures in both femurs or tibias
* Currently taking bisphosphonates
* Unable to stand independently
* Orthopedic surgery on a lower extremity within the last 6 months
* Children with pure athetoid CP
* Baclofen pump in the abdomen
* Botox treatment within the last year

Ages: 5 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Estimated)
Dates: Start 2019-01-23 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Change in fat concentration | Baseline, 6 months and 12 months
  Change in fat concentration assessed using imaging techniques

SECONDARY OUTCOMES:
Change in muscle size | Baseline, 6 months and 12 months
  Change in muscle size assessed using imaging techniques
Change in physical activity | Baseline, 1 month, 6 months, 7 months, and 12 months
  Change in physical activity assessed using activity monitors
Change in dynamic balance | Baseline, 1 month, 6 months, 7 months, and 12 months
  Change in dynamic balance assessed using step recovery method
Change in static balance | Baseline, 1 month, 6 months, 7 months, and 12 months
  Change in static balance assessed using force plates

CONTACTS AND LOCATIONS:
Overall Officials: Christopher M Modlesky, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Khan OA, Singh T, Barany DA, Modlesky CM. Accuracy deficits during robotic time-constrained reaching are related to altered prefrontal cortex activity in children with cerebral palsy. J Neuroeng Rehabil. 2024 Dec 19;21(1):216. doi: 10.1186/s12984-024-01502-x. PMID 39702205